CLINICAL TRIAL: NCT01290666
Title: Multicenter,Prospective, Observational Study of GORE® BIO-A® Fistula Plug for Use in Anal Fistula Repair
Brief Title: Study of GORE® BIO-A® Fistula Plug for Use in Anal Fistula Repair
Status: Terminated | Type: Observational
Why Stopped: Sufficient patient population achieved; decision not due to product complaints.
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: CS157
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GORE® BIO-A® Fistula Plug: All patients in study receive the GORE® BIO-A® Fistula Plug.
  Interventions: Device: Fistula Plug

INTERVENTIONS:
Device: Fistula Plug — Bioabsorbable fistula plug
  Other Names: GORE® BIO-A® Fistula Plug

SUMMARY:
Primary outcome variable is healing at the final follow up visit.

DETAILED DESCRIPTION:
The primary purpose of this prospective, multicenter, observational, single arm study is to further substantiate efficacy of the GORE® BIO-A® Fistula Plug when used as a soft tissue reinforcement of anal fistula repair and healing.

ELIGIBILITY:
Inclusion Criteria:

* Transsphincteric fistula consisting of 1 tract(defined as a fistula which would not be amenable to fistulotomy); determined during operative procedure
* Likely cryptoglandular origin
* Must be at least 18 years of age
* Patients informed about the study, and will have read, understood and signed the patient informed consent and authorization to use PHI data, as applicable
* Patients willing and able to submit to postoperative follow-up evaluations

Exclusion Criteria:

* Crohn's Disease
* Evidence of on-going local infection
* History of more than 2 prior definitive repair attempts; repair attempt is defined as any of the following: advancement flap, cutting seton, fistulotomy, fistulectomy, fibrin glue, anal fistula plug, LIFT
* Superficial fistulas without any muscle involvement
* Fistulae of traumatic origin, including obstetric
* Intersphincteric fistulas that would be candidate for fistulotomy
* Horseshoe or multi-tract fistulas
* Ano-vaginal or recto-vaginal fistulas
* Anastomotic fistulas (ileo-anal, colo-anal)
* A wound-healing or autoimmune disorder (including insulin-dependent diabetics)
* Subjects who are immunocompromised such as, with HIV, or currently receiving chemo or radiation therapy
* Subjects who are immunosuppressed, e.g. transplant patients, patients taking steroids, TNF agents, methotrexate
* History of prior or current pelvic radiation
* Difficulty comprehending or complying with the study (in surgeon's opinion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting with anal fistulae that meet inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Stamos, MD, Principal Investigator — University of California, Irvine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stamos MJ, Snyder M, Robb BW, Ky A, Singer M, Stewart DB, Sonoda T, Abcarian H. Prospective multicenter study of a synthetic bioabsorbable anal fistula plug to treat cryptoglandular transsphincteric anal fistulas. Dis Colon Rectum. 2015 Mar;58(3):344-51. doi: 10.1097/DCR.0000000000000288. PMID 25664714

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 93 subjects were recruited from 11 sites between March of 2011 and September 2013.
Period: Overall Study
Arm/Group | GORE® BIO-A® Fistula Plug
Started | 93
Completed | 55
Not Completed | 38
Not completed — Lost to Follow-up | 11
Not completed — Withdrawal by Subject | 23
Not completed — Early Termination of Study | 4

BASELINE CHARACTERISTICS:
Arm/Group | GORE® BIO-A® Fistula Plug
Number analyzed (Participants) | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 80
  >=65 years | 13
Gender [Count of Participants; unit: Participants]
  Female | 22
  Male | 71
Region of Enrollment [Number; unit: participants]
  United States | 93

OUTCOME MEASURES:

1. Primary Outcome: Fistula Closure
Time Frame: 12 months post procedure
Measure: Number; unit: participants
Arm/Group | GORE® BIO-A® Fistula Plug
Number analyzed (Participants) | 55
participants | 35

2. Secondary Outcome: Duration of Drainage Post Procedure
Time Frame: Follow up out to 12 months post procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | GORE® BIO-A® Fistula Plug
Serious Adverse Events (participants affected / at risk) | 0/93
Other Adverse Events (participants affected / at risk) | 45/93
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE® BIO-A® Fistula Plug (N=93)
Infection (Infections and infestations) | 7 (15)
Extrusion (General disorders) | 6 (16)
Unresolved Fistula (General disorders) | 7 (12)
Other (General disorders) | 25 (56)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less